CLINICAL TRIAL: NCT04966767
Title: Intermediate and Long-term Efficacy of Endovascular Treatment for TASC C&D Aortoiliac Occlusive Disease: a Prospective, Multicenter, Real-world, Registry Study
Brief Title: Intermediate and Long-term Efficacy of Endovascular Treatment for TASC C&D Aortoiliac Occlusive Disease
Acronym: ALLIANCE
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: RenJi Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Chengdu University of Traditional Chinese Medicine (Other); Xuanwu Hospital, Beijing (Other); First People's Hospital of Hangzhou (Other); Qingdao Hiser Medical Group (Other); Second Affiliated Hospital of Soochow University (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-426
Record Dates: First submitted 2021-07-09; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multicenter, real-world, registry study, which aims to observe the intermediate and long-term efficacy of different endovascular treatments for TASC C&D aortoiliac occlusive disease.

DETAILED DESCRIPTION:
Currently, the optimal therapy for TASC C and D type aortic occlusive disease is still controversial. The evidence comes from several singe-center studies with small sample size. In addition, the long-term efficacy of stent implantation and drug coated device in aortic occlusive disease remains unclear, which might be affected by the type of stent and calcification extent. Thus, this study aims to observe the intermediate and long-term efficacy of different endovascular treatments for TASC C&D aortoiliac occlusive disease in multiple centers.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford classification of 3-6
* Willing to comply with all follow-up evaluations at the specified times
* Target lesion(s) located within the native infrarenal abdominal aorta and/or common iliac artery and/or external iliac artery
* Evidence of ≥ 50% stenosis, restenosis (from PTA or adjunct therapy, not including stents or stent grafts), or occlusion of target lesion(s), or arterial thrombosis underwent PMT or CDT
* Provides written informed consent

Exclusion Criteria:

* Contraindication or known untreatable allergy to antiplatelet therapy, anticoagulants, thrombolytic drugs, or any other drug used during the study
* Known hypersensitivity to contrast material that cannot be adequately pretreated
* Bleeding diathesis or coagulopathy, known hypercoagulable condition or refuses blood transfusion
* Female currently breastfeeding, pregnant, or of childbearing potential not using adequate contraceptive measures
* Life expectancy less than 24 months
* Current participation in an investigational drug or other device study
* Severe comorbid conditions
* Myocardial infarction or stroke within 3 months prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with TASC C&D aortoiliac occlusive disease
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Free from clinically-drived target lesion reintervention | 5 years
  TLR was deﬁned as a reintervention performed for >50% diameter stenosis or in the target lesion after documentation of recurrent clinical symptoms following the index procedure or bailout stenting during the index procedure. Freedom form TLR were defined as the rates of the number of patients who did not receive reintervention verse the number of patients during the follow-up period.

SECONDARY OUTCOMES:
Technique success rate | 30 days
  Successfully revascularize the target vessel. The residual stenosis is <30% and there is no acute thrombosis occurred in the target vessel within 30 days post-operation. The Technical success rate was defined as the rate of the number of patients who receive the treatment as intended verse the number of the patients enrolled.
Perioperative adverse events | 30 days
  Perioperative adverse events include anyone of the following: all-cause mortality, Myocardial infarction, ischemic stroke, acute limb ischemia, and major amputation of a vascular etiology, and arterial thrombosis related to endovascular manipulation.
Primary patency rate | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The primary patency rate was defined as the percentage of stent patency examined by ultrasonograpy or computed tomography angiography examination of lower limb arteries during follow-up.
Incidence of adverse blood supply events | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  Incidence of adverse blood supply events include anyone of the following: acute or chronic occlusion of target lower extremity, major or minor amputation of a vascular etiology
Vascular quality of life questionnaire(VascuQol) | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
  The VascuQol was designed as a questionnaire containing five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items) to evaluate Health related quality of life (HRQL). Every item has seven response options, with scores ranging from 1 to 7. A total score is the sum of all 25 item scores divided by 25.And both the total score as well as the domain scores range from 1 (worst HRQL) to 7 (best HRQL).The lower the value, the poorer the quality of life.
Total Cost of treatment | 3 years, 5 years
  All the cost related to the target vessel and spent in the inpatient ward will be recorded and analyzed. Health economics evaluation